CLINICAL TRIAL: NCT01557426
Title: Soft Tissue Ultrasound of Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 304321
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2012-03

CONDITIONS: Soft Tissue Infections; Cellulitis; Abscess
Keywords: skin; soft tissue; infection; cellulitis; abscess
MeSH Terms: conditions — Soft Tissue Infections; Cellulitis; Abscess; Infections | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound (Other): Single interventional group - patients agree to an ultrasound of their skin or soft tissue infection and an ultrasound to an uninfected portion of skin.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — A linear ultrasound transducer will be used with ultrasound gel to obtain an image of subcutaneous structures and tissues over the involved body site. Ultrasound video will be recorded whenever possible, however studies that are not recorded will still be included. Video recording will be initiated once the desired image is obtained. Appropriate measurements will be made and views identified using the features of the ultrasound machine. Scanning of the contralateral body segment will then be performed. The ultrasound probe will be thoroughly cleaned and disinfected between ultrasound scans.

SUMMARY:
Objectives:

This study aims to characterize severe skin and soft tissue infections (SSTIs) in the emergency department through the acquisition of ultrasound images. A wide range of SSTIs will be imaged and recorded, leading to a registry of these infections. The registry will show whether ED (emergency department) sonographers can accurately characterize these infections, as compared to the final hospital diagnosis. The registry will also provide data for a case-control study comparing ultrasonographic characteristics of necrotizing skin and soft tissue infections (NSTIs) to those of non-necrotizing SSTIs.

Research procedures:

In this study, the investigators will approach patients who present to the Emergency Department with a possible skin and/or tissue infection. Study subjects must be ED patients requiring admission to the hospital for the primary problem of an SSTI due to the need for follow-up. If the patient consents to participating in the study, the investigator will obtain and record an ultrasound image of the infected area. An ultrasound image of an uninfected area of skin will also be recorded for comparison. Patient information regarding personal history, physical examination, blood tests and x-rays will also be gathered from participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand risks/benefits and consent to participation in the study
* Ability to read and understand English or Spanish
* Primary diagnosis for admission is SSTI, including cellulitis, abscess, fasciitis, myositis
* Requiring admission to an inpatient service

Exclusion Criteria:

* Patients in custody of law enforcement
* Patients on a psychiatric hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Discharge diagnosis | 2 years
  Discharge diagnosis will be collected by retrospective chart review

SECONDARY OUTCOMES:
Disposition after admission | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Otto Liebmann, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States